CLINICAL TRIAL: NCT01254487
Title: A Postmarket Surveillance Registry of the BioMatrix Drug-eluting Stent
Brief Title: e-BioMatrix PostMarket Surveillance Registry
Status: Completed | Type: Observational
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 07EU01
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the e-BioMatrix PMS registry is to capture clinical data of the BioMatrix (Biolimus A9-Eluting) stent system in relation to safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients that need a treatment with a BioMatrix™ drug-eluting stent
3. Presence of one or more coronary artery stenoses in a native coronary artery or a saphenous bypass graft from 2.25 to 4.0 mm in diameter that can be covered with one or multiple stents
4. No limitation on the number of treated lesions, and vessels, and lesion length

Exclusion Criteria:

1. Inability to provide informed consent
2. Patients needing additional stent NOT of the BioMatrix™ type
3. Patients receiving next to the BioMatrix™ stent also other coronary vascular interventions, for example dilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: "Real world, all comer" patients
Sampling Method: Non-Probability Sample
Enrollment: 1121 (Actual)
Dates: Start 2008-03; Primary Completion 2012-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) in the overall population, defined as composite of cardiac death, myocardial infarction (Q-wave and non-Q-wave), or justified target vessel revascularization | 12 Months

SECONDARY OUTCOMES:
Primary and secondary stent thrombosis (definite and probable according to ARC definitions) | 30 days, 6 and 12 months, 2, 3 and 5 years
Major adverse cardiac events (MACE) in the overall population, defined as composite of cardiac death, myocardial infarction (Q-wave and non-Q-wave), or justified target vessel revascularization | 30 days, 6 months, 2, 3 and 5 years
Patient Oriented Composite Endpoint defined as any cause mortality, MI (Q-wave and non-Q-wave), or any clinically driven target vessel revascularization | 30 days, 6 and 12 months, 2, 3 and 5 years
Death and MI | 30 days, 6 and 12 months, 2, 3 and 5 years
Total revascularization rate (clinically and non clinically driven) | 30 days, 6 and 12 months, 2, 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Philip Urban, MD, Principal Investigator — Hôpital de La Tour
Locations (9):
- Arrixaca University Hospital, Murcia, Spain
- Switzerland (6):
  - Inselspital, Bern
  - Hôpital Cantonal de Fribourg, Fribourg
  - Hôpitaux Universitaires de Genève, Geneva
  - Cardiocentro Ticino, Lugano
  - Hôpital de La Tour, Meyrin
  - Triemli Hospital, Zurich
- United Kingdom (2):
  - Brighton-Sussex University Hospitals, Brighton
  - Manchester Heart Center, Manchester